CLINICAL TRIAL: NCT03090490
Title: Clinical Outcome After Antipsychotic Treatment Discontinuation in Functionally Recovered First-episode Non-affective Psychosis Individuals: a 10-year Follow-up
Brief Title: 10-year Follow-up of Clinical Outcome After Antipsychotic Treatment Discontinuation in Psychosis Individuals
Acronym: ADARFEP_10Y
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADARFEP_10Y
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia; Schizophrenia Relapse; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Treatment; Maintenance
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Antipsychotic treatment discontinuation (DT)
  Interventions: Other: Antipsychotic treatment discontinuation
- Control group (Active Comparator): Maintenance antipsychotic treatment (MT)
  Interventions: Other: Maintenance treatment discontinuation

INTERVENTIONS:
Other: Antipsychotic treatment discontinuation — Withdrawal of antipsychotic medication to stabilized patients
  Arms: Intervention group
Other: Maintenance treatment discontinuation — Maintenance antipsychotic medication to stabilized patients
  Arms: Control group

SUMMARY:
This open-label, non-randomized, prospective study will evaluate the risk of symptoms recurrence during the ten years after antipsychotic discontinuation in a sample of functionally recovered first-episode patients with schizophrenia spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander, Spain).
* A minimum of 18 months on antipsychotic treatment.
* Meeting clinical remission criteria for at least the 12 months prior to inclusion.
* Meeting the functional recovery criteria for at least the 6 months prior to inclusion.
* Stabilized at the lowest effective doses for at least the 3 months prior to inclusion.

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | At 10 years
  The percentage of relapse/exacerbation in the two groups of patients, discontinuation and maintenance.

SECONDARY OUTCOMES:
Change in general psychopathology measured by BPRS | At 10 years
  Measured by changes in total score of the Brief Psychiatric Rating Scale (BPRS).
Change in overall clinical status measured by CGI | At 10 years
  Measured by changes in total score of the Clinical Global Impression (CGI).
Change in negative symptoms measured by SANS | At 10 years
  Measured by changes in total score of the Scale for the Assessment of Negative Symptoms (SANS).
Change in negative symptoms measured by SAPS | At 10 years
  Measured by changes in total score of the Scale for the Assessment of Positive Symptoms (SAPS).
Time to relapse | At 10 years
  Time to relapse in the two groups of patients, discontinuation and maintenance.
Functionality status measured by DAS | At 10 years
  Measured by changes in total score of the Disability Assessment Scale (DAS).

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No